CLINICAL TRIAL: NCT05643937
Title: Construction and Application of Precise Health Education Model for Patients With PICC Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junyan Zhao (Other)
Responsible Party: Sponsor-Investigator, Junyan Zhao, Principal investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YXLL-KY-2022(067)
Record Dates: First submitted 2022-08-24; First posted 2022-12-09 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Tumor Chemotherapy Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Active Comparator): The control group received routine health education after catheterization, including introducing the purpose, method, advantages and complications of PICC insertion to patients before catheterization and signing informed consent. During catheterization, PICC assistant explained relevant matters needing attention and cooperative actions to the patient. After catheterization, patients were instructed to carry out grip training and limb activities.
  Interventions: Behavioral: Routine health education
- Experimental group (Experimental): On the basis of routine health education in the control group, the experimental group screened the high-risk behaviors of patients through the questionnaire of daily life behavior habits, and formulated the precise and concrete health education program for their high-risk behaviors
  Interventions: Behavioral: Routine health education + precise health education

INTERVENTIONS:
Behavioral: Routine health education — The control group received routine health education after catheterization, including introducing the purpose, method, advantages and complications of PICC insertion to patients before catheterization and signing informed consent. During catheterization, PICC assistant explained relevant matters needing attention and cooperative actions to the patient. After catheterization, patients were instructed to carry out grip training and limb activities.
  Arms: The control group
Behavioral: Routine health education + precise health education — On the basis of routine health education in the control group, the experimental group screened the high-risk behaviors of patients through the questionnaire of daily life behavior habits, and formulated the precise and concrete health education program for their high-risk behaviors
  Arms: Experimental group

SUMMARY:
1. In this study, the risk factors leading to catheter-related complications in the daily life behavior habits of patients with PICC catheter were identified, refined and initially established, and the Delphi method (expert consultation method) was used to further identify the existing and potential risk factors leading to PICC catheter-related complications in the daily life behavior habits of patients. To develop individualized and precise health education programs for risk factors, in order to build an accurate health education model centered on improving patients' daily life and behavior habits.
2. To conduct clinical empirical study to evaluate the feasibility and effectiveness of precise health education program for PICC patients with catheter, and to observe the impact of this health education model on the knowledge, attitude and practice level of daily management, self-management efficacy and the incidence of related complications after catheter insertion in PICC patients, so as to provide a reference for health education of PICC patients.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients undergoing chemotherapy in our hospital with ≥6 cycles of chemotherapy;
* Patients with PICC implanted for the first time and maintained at our hospital;
* Aged 18-60 years;
* The material and performance of PICC catheter are silicone three-way valve catheter;
* Catheter placement under the guidance of portable color Doppler ultrasound diagnostic instrument;
* Clear consciousness, good language communication skills and normal comprehension ability;
* Informed consent and voluntary participation in the study.

Exclusion Criteria:

* Persons with self-care ability defects;
* Puncture times more than 1 time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of complications associated with PICC catheter | Six cycles of chemotherapy,Each chemotherapy cycle lasted 28 days
  It is determined by PICC specialist nurse/sonographer during each patient maintenance

SECONDARY OUTCOMES:
Knowledge, attitude and practice score of daily management of patients with PICC tube | Patients before catheterization and after 6 cycles of chemotherapy
  Through the results of PICC daily management knowledge, attitude and practice questionnaire, the scores of daily management knowledge, attitude and practice before and after intervention were analyzed and compared between the two groups
Scores of self-management efficacy of patients with PICC tube | A total of 6 chemotherapy cycles were observed before catheterization and after each chemotherapy cycle (28 days)
  Through the results of self-management efficacy questionnaire of patients with PICC tube, the scores of self-management efficacy before and after intervention were analyzed and compared between the two groups.
Satisfaction of health education of patients with PICC tube | A total of 6 chemotherapy cycles were observed before catheterization and after each chemotherapy cycle (28 days)
  Through the results of the health education satisfaction questionnaire of patients with PICC tube, the satisfaction of the two groups of patients with health education after intervention was analyzed and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided